CLINICAL TRIAL: NCT03288961
Title: Development and Validation of Patient Self-screening and Monitoring Tool for Crohn's Perianal Fistula
Brief Title: Self Screening Tool for Crohn's Perianal Fistula
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Associate professor, Kyungpook National University Hospital
Other Study IDs: KNUH14
Record Dates: First submitted 2017-09-19; First posted 2017-09-20 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a self-screening tool for Crohn's perianal fistula.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease

Exclusion Criteria:

-

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Crohn's disease patients are asked to fill out survey of their perianal symptoms. Survey score is compared with MRI results as the gold standard.
Sampling Method: Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Perianal fistula | 1 day
  perianal fistula rate confirmed by MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea